CLINICAL TRIAL: NCT02328638
Title: Development of a Manual-based, Interdisciplinary Intervention for Youth With ASD and Obesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Kristen K. Criado, Kristen Criado, Ph.D., Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00073170
Record Dates: First submitted 2014-12-23; First posted 2014-12-31 (Estimated); Last update posted 2016-01-20 (Estimated); Status verified 2016-01

CONDITIONS: Autism; Obesity
Keywords: ASD
MeSH Terms: conditions — Autistic Disorder; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Manual-based Behavioral Treatment (Active Comparator): up to 16 weekly behavioral therapy sessions (intervention) following the CHANGE obesity manual, lasting approximately 45 minutes and nutritional therapy sessions, lasting approximately 30 to 60 minutes.
  Interventions: Behavioral: Manual-based Behavioral Treatment
- Parent Education Program (Placebo Comparator): up to 16 weekly behavioral therapy sessions following the parent education program
  Interventions: Behavioral: Parent Education Program

INTERVENTIONS:
Behavioral: Parent Education Program — The PEP intervention consists of didactic sessions regarding basic information about Autism Spectrum Disorders.
  Other Names: PEP
  Arms: Parent Education Program
Behavioral: Manual-based Behavioral Treatment — The Manual-based Interdisciplinary Behavioral Treatment consists of nutritional and behavioral interventions to improve dietary intake (increase water, decrease sweetened beverages and snack foods, improve balanced diet), increase exercise, and teach behavioral strategies to address barriers to these goals.
  Arms: Manual-based Behavioral Treatment

SUMMARY:
The purpose of the proposed study is to develop and pilot test a manual-based, interdisciplinary intervention for youth, ages 3 to 10 years, with autism spectrum disorder (ASD) and overweight called the Changing Health in Autism through Nutrition, Getting fit, and Expanding variety (CHANGE) obesity program.

DETAILED DESCRIPTION:
The purpose of the study is to develop and test the feasibility of a structured, innovative approach to treat obesity in 16 children (age 3 to 10 years) with autism spectrum disorder (ASD). This 16-week program integrates behavioral psychology and nutrition science to meet the challenges of obesity in children with autism spectrum disorder (ASD). The PI will apply an evidence-based behavioral intervention to increase food variety,15 use applied behavior analytic strategies to teach physical activities in a developmentally-appropriate manner, employ biometrics to assess progress, utilize dietetic interventions to improve nutritional balance, and train caregivers to use behavior management strategies.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of ASD confirmed by a clinical psychologist using a "gold standard" diagnostic tools
* Overweight status, as evidenced by a BMI percentile > 85% to 94%, and 4) mild to no food selectivity, as evidenced by either history of consuming some fruits and vegetable, tolerating new foods near their plate, and/or trying new foods

Exclusion Criteria:

* Children being treated with atypical antipsychotics (e.g., olanzapine, aripiprazole, risperidone) or other medications known to cause weight gain will be excluded from the study due to the weight gain associated with these medications
* Children with unstable medical conditions will be excluded for safety concerns
* Children presenting with severe aggression, self injury, or other disruptive behaviors that require intensive behavioral intervention will be excluded and referred to other services as needed

Ages: 3 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Actual)
Dates: Start 2014-12; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Change in body mass index percentile/ratio | baseline, post treatment (up to 16 weeks)
  Body Mass Index (BMI) is a number calculated from a person's weight divided by height.

SECONDARY OUTCOMES:
Change in intake of healthy food | baseline, post treatment (up to 16 weeks)
  The Nutrition arm of the intervention is based on our dietitian's unique ASD-specific adaptations to Best Practices in dietetics and will be supplemented by Children's Healthcare of Atlanta's Strong4Life program.
Change in physical activity | baseline, post treatment (up to 16 weeks)
  The F.I.T.T. Principle will be applied to the physical activity recommendations by identifying the frequency, intensity, time, and type of exercise.

CONTACTS AND LOCATIONS:
Overall Officials: Kristen K Criado, Ph.D., Principal Investigator — Emory University
Locations (1):
- Pediatric Feeding Disorders Program at the Marcus Autism Center, Atlanta, Georgia, United States